CLINICAL TRIAL: NCT00950079
Title: Preventive Strategies of REnal Insufficiency in Patients With Diabetes Undergoing InterVENTion or Arteriography(PREVENT Trial)
Brief Title: Prevention of Contrast-Induced Nephropathy in Diabetic Patients With Undergoing Coronary Angiography
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Seong-Wook Park, MD, PhD, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007-0180
Record Dates: First submitted 2009-07-06; First posted 2009-07-31 (Estimated); Last update posted 2009-07-31 (Estimated); Status verified 2009-07

CONDITIONS: Contrast Induced Nephropathy
Keywords: sodium bicarbonate; diabetes mellitus; coronary angiography or intervention
MeSH Terms: conditions — Diabetes Mellitus | interventions — Sodium Bicarbonate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium bicarbonate (Experimental): sodium bicarbonate
  Interventions: Drug: Sodium bicarbonate
- Saline (Active Comparator): saline infusion
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Sodium bicarbonate — 3 mL/kg for 1 hour immediately before contrast injection , 1mg/kg/hr during procedure and 6 hours after procedure
  Arms: Sodium bicarbonate
Drug: saline — 0.9% normal saline with 1 mL/kg/hr infusion 12 hours before procedure and 12 hours after procedure
  Arms: Saline

SUMMARY:
The aim of this study is to determine whether sodium bicarbonate is superior to sodium chloride in preventing contrast induced nephropathy in diabetic patients undergoing coronary angiography or intervention.

DETAILED DESCRIPTION:
Contrast induced nephropathy (CIN) is a common cause of renal failure associated with prolonged hospitalization, significant morbidity or mortality, and cost. CIN has been reported to account for 10% of hospital acquired renal failure. Several strategies or medications were tried to prevent CIN. Of these, mucomyst and normal saline infusion are effective to prevent CIN. Sodium bicarbonate has shown mixed results from recent randomized trials. Moreover,limited data have been available for preventing CIN in diabetic renal dysfunction undergoing coronary angiography or intervention. Our hypothesis is that addition of sodium bicarbonate will be more efficacious than normal saline in preventing CIN at above situation.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years, no upper limits
* diabetes treated with insulin or oral hypoglycemic agents
* serum creatinine >=1.1 and
* resting estimated glomerular filtration rate <60ml/min/1.73 square meter

Exclusion Criteria:

* serum creatinine >=8mg/dL
* resting estimated GFR <15ml/min/1.73 square meter
* end stage renal disease on hemodialysis
* multiple myeloma
* uncontrolled hypertension (systolic BP >160mmHg or diastolic BP>100mmHg)
* acute myocardial infarction
* emergent coronary angioplasty or angiography
* recent use of contrast within 2 days
* allergic reaction to contrast
* pregnancy
* allergic to following medication : theophylline, dopamine, mannitol, fenoldopam, N-acetylcysteine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-08 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of contrast-induced nephropathy | 24 and 48 hours after angiography or intervention

SECONDARY OUTCOMES:
all-cause mortality | 30 days after index angiography
stroke | 30 days after index angiography
Dialysis | 30 days after index angiography
Myocardial infarction | 30 days after index angiography
all-cause mortality | 30 days to 6 months after index angiography
stroke | 30 days to 6 months after index angiography
dialysis | 30 days to 6 months after index angiography
myocardial infarction | 30 days to 6 months after index angiography

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Wook Park, MD, PhD, Principal Investigator — Department of Medicine, Asan Medical Center, University of Ulsan College of Medicine
Locations (9):
- South Korea (9):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Busan Saint Mary Hospital, Busan
  - Soonchunhyang University Hospital, Cheonan, Cheonan
  - Kangwon National University Hospital, Chuncheon
  - Chungnam National University Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Asan Medical Center, Seoul
  - Soonchunhyang University Seoul Hospital, Seoul
  - Ulsan University Hospital, Ulsan